CLINICAL TRIAL: NCT03827057
Title: RECONsolidation of Traumatic Memories to ResOLve Post Traumatic Stress Disorder (RECONTROLPTSD)
Acronym: RECONTROLPTSD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: Research and Recognition Project (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNRM-83-9763
Record Dates: First submitted 2019-01-04; First posted 2019-02-01 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Posttraumatic Stress Disorder; Traumatic Brain Injury
Keywords: posttraumatic stress disorder; traumatic brain injury; cognitive behavioral therapy; exposure therapy; reconsolidation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: This is an interventional randomized controlled trial in which participants have an equal chance of receiving either the current best-evidenced PTSD treatment, prolonged exposure, or a novel approach, reconsolidation of traumatic memories, that has the potential to achieve a more rapid, durable and greater overall response rate.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The CAPS-5, the gold standard for PTSD diagnosis, will be administered and scored at baseline to confirm the diagnosis, and subsequently as the primary outcome measure at 2, 6, and 12 months, by expert administrators who will be blinded to treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reconsolidation of Traumatic Memories (RTM) (Experimental): Participants in each arm of the study will receive up to 10 90-minute manualized treatment sessions. RTM will follow a manual developed by the Research and Recognition Project, who will also train and supervise the therapists. It is anticipated that these treatments will most often be administered once per week for 10 weeks. To best meet participant needs, we will allow therapy in either arm to be "massed" in the pattern recently reported by Foa et al. for PE, with sessions separated by at least 24 hours over two weeks. This schedule has been used with both RTM and PE without hurting response rates, and may reduce drop-out rates. Participants who achieve remission of their PTSD before 10 sessions, measured by a PCL5 <34, can decide with their therapist whether early cessation of therapy is appropriate.
  Interventions: Behavioral: Reconsolidation of Traumatic Memories (RTM)
- Prolonged Exposure (PE) (Active Comparator): Participants in each arm of the study will receive up to 10 90-minute manualized treatment sessions. PE will follow a manual written by the Foa and colleagues, and the therapists will be trained by expert trainers from the Center for Deployment Psychology. It is anticipated that these treatments will most often be administered once per week for 10 weeks. To best meet participant needs, we will allow therapy in either arm to be "massed" in the pattern recently reported by Foa et al. for PE, with sessions separated by at least 24 hours over two weeks. This schedule has been used with both RTM and PE without hurting response rates, and may reduce drop-out rates. Participants who achieve remission of their PTSD before 10 sessions, measured by a PCL5 <34, can decide with their therapist whether early cessation of therapy is appropriate.
  Interventions: Behavioral: Prolonged Exposure (PE)

INTERVENTIONS:
Behavioral: Reconsolidation of Traumatic Memories (RTM) — RTM is a trauma-focused, but not cognitive behavioral, therapy: it involves brief exposure to the trauma memory, but does rely on conscious responses to correct the symptoms of PTSD. RTM was first used to treat phobias in the 1970s, and has more recently been refined to focus on reconsolidation to update long-term memories, reconfiguring the salience structure of the original memory, and incorporating those changes into the overall memory structure. Reconsolidation is a neural mechanism for updating long-term memory, inserting new information that contradicts an essential element of the memory, which makes it possible to change the emotional tone and salience of the memory. It is hypothesized that RTM can thereby achieve quicker, greater, and more durable responses than with "traditional" exposure therapies.
  Arms: Reconsolidation of Traumatic Memories (RTM)
Behavioral: Prolonged Exposure (PE) — PE is a trauma-focused cognitive behavioral therapy (TFCBT) that depends on exposure to the feared stimulus as a central effector of change, utilizing extinction, which theorizes that if a trigger that previously elicited a fear response is presented enough times without reinforcement, the response fades. Previous researchers have shown that extinction involves the creation of a new blocking memory which prevents expression of the original fear memory. While PE has more evidence to support its efficacy in PTSD than other approaches, and a majority achieve a clinical response (e.g., decrease in CAPS score of 10 or more), many do not achieve complete remission of symptoms, and the blocking memory may be fragile, so subsequent triggers may result in relapse.
  Arms: Prolonged Exposure (PE)

SUMMARY:
Posttraumatic Stress Disorder (PTSD) is a common cause of morbidity in combat veterans, but current treatments are often inadequate. Reconsolidation of Traumatic Memories (RTM) is a novel treatment that seeks to alter key aspects of the target memory (e.g., color, clarity, speed, distance, perspective) to make it less impactful, and reduce nightmares, flashbacks, and other features of PTSD. The memory is reviewed in the context of an imaginal movie theater, presenting a fast (~45 sec) black and white movie of the trauma memory, with further adjustment as needed so the patient can comfortably watch it. Open and waitlist studies of RTM have reported high response rates and rapid remission, setting the stage for this randomized, controlled, single-blind trial comparing RTM versus prolonged exposure (PE), the PTSD therapy with the strongest current evidence base.

The investigators hypothesize that RTM will be non-inferior to PE in reducing PTSD symptom severity post-treatment and at 1-year follow up; will achieve faster remission, with fewer dropouts; will improve cognitive function; and that epigenetic markers will correlate with treatment response. The investigators will randomize 108 active or retired service members (SMs) with PTSD to ≤10 sessions of RTM or PE, affording power to test our hypotheses while allowing for ≤ 25% dropouts. The investigators will use an intent to treat analysis, and the Clinician Administered PTSD Scale for the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition, or DSM5 (CAPS-5), conducted by blinded assessors, will be the primary outcome measure. Secondary measures of depression (PHQ-9), anxiety (GAD-7), sleep (PSQI), and functional status (WHOQOL-100), will be assessed pre- and post-treatment, and at 2, 6, and 12 months. ANOVA will compare symptom severity over time within and between groups. The investigators will track comorbid TBI, anticipating it will not adversely impact response. More effective therapies for PTSD, with and without TBI, must be developed and evaluated. RTM is safe and promising, but requires testing against evidence-based interventions in well-designed randomized clinical trials (RCTs). The full study can be conducted either in person or via secure video conferencing.

DETAILED DESCRIPTION:
Primary Objective: The primary intent of this study is to determine whether Reconsolidation of Traumatic Memories (RTM) achieves a greater and/or more rapid response than prolonged exposure (PE) in the treatment of military service members with PTSD. This is an interventional randomized controlled trial in which all participants will receive active psychotherapy for PTSD, either what is currently considered the best-evidenced treatment, prolonged exposure, or a novel approach, reconsolidation of traumatic memories, that the investigators believe can achieve a higher response rate that will also prove more rapid and more durable. Participants will be active duty, reserve or National Guard service members, or former service members who were retired either medically or for length of service, who are eligible for care in the Department of Defense Healthcare System. Our findings should be generalizable to current and former military service members with PTSD.

Approach This is a randomized controlled trial, enrolling 108 SMs with active PTSD, to RTM and PE, with up to 10 treatment sessions in each arm. The anticipated average enrollment rate will be 2 new participants per week. Participants may be male and female adult (ages 18+) participants who are active, reserve component, National Guard, or retired SMs; those with active suicidal or homicidal ideation, or a history of a psychotic disorder, will be excluded. Participants may have a history of lifetime mild or moderate traumatic brain injury (TBI), or no TBI history, but no lifetime history of severe TBI. Given that most participants are expected to be referred from the Center for Neuroscience and Regenerative Medicine (CNRM)'s Military Recruitment Protocol, it is anticipated that the great majority will have comorbid mild TBI (mTBI). All participants will also complete a total of 5 assessment visits: at baseline, immediately after the course of treatment, and at 2, 6 and 12 months. The baseline visit will begin with the completion of informed consent, followed by the administration of a series of questionnaires, a detailed neurocognitive assessment, and a blood draw; serial assessment will occur throughout the intervention period and for 12 months of follow-up. Participants will be randomly assigned to PE or RTM using a random number generator in MS Excel or other program to generate a random sequence of 108 zeroes and ones as a list. Subjects will be assigned to the treatment arms from that list: all zeros will be assigned to RTM and ones to PE.

Hypotheses: Military service members with PTSD who are randomized to Reconsolidation of Traumatic Memories (RTM) therapy will be significantly more likely to achieve PTSD resolution than those randomized to Prolonged Exposure (PE) therapy, measured by the Clinician-Administered PTSD Scale for DSM5 (CAPS-5, by expert assessors blinded to treatment group assignment). The investigators also anticipate that RTM will achieve a response more rapidly, and will prove more durable. Among the secondary measures that will correlate with response to therapy are measures of depression, anxiety, sleep quality, and overall functional status. Primary Aim: Compare response rates of PTSD to RTM vs. PE, defined by remission of diagnosis on the CAPS-5, using a 2-tailed t-test, from baseline to post-intervention. The investigators will also utilize repeated measures ANOVA to compare CAPS-5 scores at baseline, post-intervention, and at 2-, 6-, and 12-month follow up within groups. In addition to this primary measure, the investigators will also use independent sample t-tests to document the efficacy of randomization by comparing the two groups' baseline CAPS-5 total scores, along with PCL5, PHQ-9, NSI, GAD-7, PSQI, WHOQOL-10, number of TBIs, and all other demographic variables.

Secondary Aim 1: Corroborate impact on PTSD symptom severity by measuring changes in CAPS-5 and PCL5, respectively, from baseline to post-treatment for RTM and PE, using a 2-tailed t-test. The investigators will then use repeated measures ANOVA to compare within and between group changes in the CAPS-5 at baseline, post-treatment, 2-, 6-, and 12-month follow-up for the CAPS-5, and these as well as scores obtained prior to treatment sessions 2, 4, 6, 8 and 10 for the PCL5.

Secondary Aim 2: Compare rapidity of improvement in PTSD symptom severity between RTM and PE, measured by PCL5 scores at baseline, prior to treatment sessions 2, 4, 6, 8 and 10, and post-treatment, using a log-rank test to compare Kaplan-Meier curves for two groups.

Secondary Aim 3: Compare the durability of response to treatment, with the primary measure being the percentage meeting criteria for PTSD on the CAPS-5, at post-treatment, and at 2-, 6-, and 12-month follow-ups, using repeated measures ANOVA between the two groups. The investigators will also determine whether this is corroborated by symptom severity reduction by comparing the CAPS-5 and PCL5 scores at these time points, again using repeated measures ANOVA.

Secondary Aim 4: Compare the impact of RTM and PE upon comorbid conditions by using ANOVA with Bonferroni adjustment for multiple comparisons, to compare scores at baseline, post-treatment, and each of the follow-up time-points, on postconcussive symptoms (NSl), depression (PHQ-9), anxiety (GAD-7), sleep (PSQI), and functional status (WHOQOL-100).

ELIGIBILITY:
Inclusion Criteria:

1. Meets criteria for PTSD on the CAPS5, with past month nightmares or flashbacks.
2. Willing to be randomly assigned to one of the two interventions and to complete all study measures.
3. Able to exhibit capacity to understand the informed consent process, by completion of a corresponding series of questions

Exclusion Criteria:

1. history of psychosis, bipolar disorder, or active suicidal or homicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Symptom Scale for DSM5 (CAPS-5) | week 10
  the gold standard for PTSD diagnosis, a trained expert administrator scores PTSD symptom severity; range 0-80, higher score represents greater severity

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire (PHQ-9) Score | week 10, and 2, 6 and 12 months later, compared to baseline
  well-validated and widely used 9-item self-report measure of depression symptom severity, range 0-27, higher score represents greater severity
Change in PTSD Checklist for DSM5 (PCL5) Score | week 10, and 2, 6 and 12 months later, compared to baseline
  a reliable 20-item screen for PTSD, in which each item is rated on a 5-point Likert scale, range 0-80, higher score represents greater severity
Change in Pittsburgh Sleep Quality Index (PSQI) Score | week 10, and 2, 6 and 12 months later, compared to baseline
  a clinically validated 9-item assessment of sleep quality and sleep disturbances; range 0 to 21, higher score represents greater severity
Change in Neurobehavioral Symptom Inventory (NSI) Score | week 10, and 2, 6 and 12 months later, compared to baseline
  a reliable 22-item self-report measure assessing functional status and post concussive symptoms, range 0-88, higher score represents greater severity
Change in World Health Organization Quality of Life Inventory (WHOQOL-100) Score | week 10, and 2, 6 and 12 months later, compared to baseline
  a reliable 100 item self-report inventory measuring overall quality of life in 8 dimensions; range 100 to 500, higher score represents greater severity

CONTACTS AND LOCATIONS:
Locations (1):
- Uniformed Services University of Health Sciences (USUHS), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be entered into the Federal Interagency TBI Research Informatics System (FITBIR) through the CNRM after completion of the study and after all codes or links to personal identifying information have been destroyed.
Supporting Information: CSR
Time Frame: after study completion
Access Criteria: Must have approved research protocol
URL: https://fitbir.nih.gov/

DOCUMENTS (1):
  • Informed Consent Form (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/57/NCT03827057/ICF_000.pdf